CLINICAL TRIAL: NCT03007615
Title: Dermal and Gynecological Acceptability (Irritability and Sensitization in the Genital Mucosa) of an Investigational Product and Evaluation of Moisture Efficacy by TEWL and Perceived Efficacy.
Acronym: DERM GYN ACCEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kley Hertz S/A (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: Kley Hertz 007
Record Dates: First submitted 2016-12-29; First posted 2017-01-02 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-12

CONDITIONS: Female Dry Genital Mucosa

STUDY DESIGN:
Who Masked: Participant

ARMS (1):
- Experimental group (Experimental)
  Interventions: Other: Intimate Lubricant Gel

INTERVENTIONS:
Other: Intimate Lubricant Gel

SUMMARY:
To evaluate the safety of an investigational product through the verification of signs of irritability and sensitization of the genital mucosa, as well as the instrumental moisturizing efficacy by TEWL and barrier integrity analysis, in addition to the efficacy perceived by the volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female sex with active sex life;
* Age group: between 45 and 65 years old;
* Menopause for at least six months;
* Whole skin in the region of product analysis;
* No history of reaction to products of the same category
* Understanding, agreement and signature of the Term of Free and Informed Consent.

Exclusion Criteria:

* Gestation or risk of gestation;
* Use of anti-inflammatory / immunosuppressive drugs (in the last 30 days and during the study);
* Active cutaneous pathologies (local and / or disseminated) in the evaluation area;
* Pathologies that cause suppression of immunity, such as diabetes, HIV, etc.;
* Endocrine pathologies such as thyroid disorders, ovarian or adrenal gland disorders;
* Any infection in the region of analysis of the product diagnosed at the time of inclusion;
* Other conditions considered by the investigating physician as reasonable for disqualification of the individual from the study participation.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the product's efficiency as a moisturizer through subjective evaluation | 30 days